CLINICAL TRIAL: NCT03933033
Title: Fractional Erbium-YAG Laser Versus Platelet Rich Plasma in the Treatment of Atrophic Acne Scars: A Randomized Clinical Trial
Brief Title: Erbium-YAG Laser Versus Platelet Rich Plasma in the Treatment of Atrophic Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Collaborators: South Valley University (Other)
Responsible Party: Principal Investigator, Moustafa A. El Taieb, Ass. Prof. of Dermatology, Venereology and Andrology, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Erbium Yag
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Acne Vulgaris; Scars
Keywords: Acne scars; Erbium-YAG laser; platelet-rich plasma
MeSH Terms: conditions — Acne Vulgaris; Cicatrix

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): treated with platelet rich plasma
  Interventions: Procedure: Platelet Rich Plasma
- Group B (Active Comparator): treated with Erbium Yag Laser
  Interventions: Device: Fractional Erbium Yağ Laser
- Group C (Active Comparator): treated with both line of treatments
  Interventions: Device: Fractional Erbium Yağ Laser; Procedure: Platelet Rich Plasma

INTERVENTIONS:
Device: Fractional Erbium Yağ Laser — Multiple sessions of Fractional Erbium Yağ Laser
  Arms: Group B; Group C
Procedure: Platelet Rich Plasma — Multiple injections of Platelet Rich Plasma
  Arms: Group A; Group C

SUMMARY:
This study aim to assess the efficacy of Er-YAG laser 2940nm and PRP as a single line of treatment in comparison with combined treatment in atrophic post acne scars.

ELIGIBILITY:
Inclusion Criteria:

* patients with atrophic post acne scars classified on the basis of Goodman and Baron's Qualitative classification, no active acne lesions and patients with atrophic scars only

Exclusion Criteria:

* patients with positive history of keloidal tendency, positive history of bleeding tendency, platelet disorder, patients with any acute infection on face like, herpes, folliculitis, patients with HIV, HBsAg, patients with a history of autoimmune diseases or patients on immunosuppressive drugs.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in grade of acne scares according toQualitative scarring grading system of Goodman and Baron | 6 months
  Grade of acne scares improvement after treatment
Change in clinical appearance of acne scare accordinga four-point scale for assessment of clinical improvement of skin smoothness | 6 month
  improvement of acne scares as evaluated by sequential photos
Change in patient satisfaction usinga four-point scale; Grade 4 highly satisfied, Grade 3 satisfied, Grade 2 neutral and Grade 1 dissatisfied | 6 month
  increase in patient satisfaction after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Taieb MA, Ibrahim HM, Hegazy EM, Ibrahim AK, Gamal AM, Nada EA. Fractional Erbium-YAG Laser and Platelet-Rich Plasma as Single or Combined Treatment for Atrophic Acne Scars: A Randomized Clinical Trial. Dermatol Ther (Heidelb). 2019 Dec;9(4):707-717. doi: 10.1007/s13555-019-00318-1. Epub 2019 Aug 16. PMID 31420849